CLINICAL TRIAL: NCT03829592
Title: TheEffect of pH on Misoprostol in Induction of Labor in Full Term Pregnancies
Brief Title: TheEffect of pH on Misoprostol in Induction of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Misoprostol
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Misoprostol; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: 3 paralle groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- misoprostol in neutral media (Placebo Comparator): Intervention : misoprostol in a neutral media will be given to women to induce labour
  Interventions: Drug: misoprostol in a neutral media
- Misoprostol in acidic media (Active Comparator): Intervention : misoprostol in acidic media will be given to induce labour
  Interventions: Drug: misoprostol in an acidic media
- Misoprostol in alkaline media (Sham Comparator): Intervention : misoprostol in alkaline media will be given to induce labour
  Interventions: Drug: misoprostol in an alkaline media

INTERVENTIONS:
Drug: misoprostol in a neutral media — giving misoprostol in a neutral media
  Other Names: Drug (misoprostol + neutral media )
  Arms: misoprostol in neutral media
Drug: misoprostol in an acidic media — giving misoprostol in an acidic media
  Other Names: Drug ( Misoprostol + acidic media )
  Arms: Misoprostol in acidic media
Drug: misoprostol in an alkaline media — giving misoprostol in an alkaline media
  Other Names: Drug ( misoprostol + alkaline media )
  Arms: Misoprostol in alkaline media

SUMMARY:
Misoprostol is a synthetic analogue of the naturally occurring prostaglandin E1. It was initially marketed for the treatment of peptic ulcers due to its mucosal protective and anti-secretory properties, but has commonly been used for the induction of abortion and labour .

DETAILED DESCRIPTION:
Although initially having been established for oral use, misoprostol tablets are commonly used as vaginal suppositories for the previously purposes. Water or saline are frequently used in common practice to moisten the tablets prior to their administration, however, according to the pharmacokinetics of the drug, it should liquefy better in an acidic medium

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies. Gestational age 38-41 weeks. Cephalic presentation

Exclusion Criteria:

* 1. Multi-fetal pregnancy. 2. Pregnant women less than 38 weeks gestation.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Full term pregnant women
Enrollment: 180 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-07-12 (Estimated)

PRIMARY OUTCOMES:
The number of women who will start lactive phase of labour after treatment | within 24 hours
  the number of women in a group who will enter in active labour faster than other groups

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt